CLINICAL TRIAL: NCT05468463
Title: Promoting Increases in Living Donation Via Tele-navigation (PILOT)
Acronym: PILOT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Vineeta Kumar, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-300002556; R01DK125509 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Kidney Diseases
Keywords: Kidney Disease; Kidney; End Stage Kidney Disease; Living Donation; Telehealth; Transplant; Remote; Virtual
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living Donor Navigator Program In-person (Active Comparator): The LDN program is designed to help transplant candidates find potential donors, and guide potential living donors through the evaluation/ donation process. The LDN program consists of four educational sessions, with each session building on the last. Each educational session lasts approximately 2 hours and is held once every other week for two months. Each LDN session will be conducted by a living donor navigator. As potential living donors are identified, the living donor navigators will work closely with the potential donors to guide them through each step of the evaluation/donation process to ensure streamlined medical services and a personalized experience. Individuals randomized to LDN in-person will receive the program locally at the transplant center.
  Interventions: Behavioral: Living Donor Navigator Program
- Living Donor Navigator Program Tele-health (Active Comparator): The LDN program is designed to help transplant candidates find potential donors, and guide potential living donors through the evaluation/ donation process. The LDN program consists of four educational sessions, with each session building on the last. Each educational session lasts approximately 2 hours and is held once every other week for two months. Each LDN session will be conducted by a living donor navigator. As potential living donors are identified, the living donor navigators will work closely with the potential donors to guide them through each step of the evaluation/donation process to ensure streamlined medical services and a personalized experience. Individuals randomized to LDN tele-health will receive the program virtually at a local health department within the Alabama Department of Public Health's tele-health network.
  Interventions: Behavioral: Living Donor Navigator Program

INTERVENTIONS:
Behavioral: Living Donor Navigator Program — The investigators have developed a 4-session educational program that simultaneously addresses potential donor concerns with the evaluation/donation process and provides advocacy training to transplant candidates and their advocates.

SUMMARY:
We hypothesize that expansion of the Living Donor Navigator (LDN) program to include tele-health delivery will overcome geographic disparities in access and facilitate sustained increases in living donation. We will utilize an individually randomized group trial (IRGT) design with delayed intervention initiation to compare the effectiveness of tele-health LDN model to standard of care.

DETAILED DESCRIPTION:
Transplant candidate-related and potential living donor-related factors, including difficulty asking family/friends to donate on one's behalf and lack of knowledge about the donation process, respectively, have been implicated in lower donation rates. The investigators will conduct an individually randomized group trial (IRGT) with delayed intervention initiation allowing for: (1) scalability/ implementation in a less resource-intensive fashion compared to traditional randomized trials; (2) Avoid self-selection bias as all participants ultimately participate in the intervention. The LDN Program combines advocacy-training to overcome barriers in initiating conversations with and identification of potential living donors with the use of non-clinical navigators to guide donors through the evaluation process. Participants will be randomized to one of two arms; Arm 1 includes the LDN program via in-person modality, and Arm 2 includes the LDN program via tele-health modality. The investigators primary objective is to demonstrate the effectiveness of these interventions in increasing living donation.

ELIGIBILITY:
Inclusion Criteria:

* End-stage kidney disease (ESKD) patients who are ≥ 18 years old and have initiated evaluation for kidney transplantation.
* If there is an individual willing to donate, but the candidate is unwilling to consider this option or this particular individual, the candidate is eligible for the study and may still benefit from identification of new donors or increased comfort accepting donation from others.
* Candidates must be English-speaking or deaf with an interpreter.

Exclusion Criteria:

* Individuals under the age of 18 will be excluded from the study.
* Individuals who are not English speaking will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number Live Donor Screenings | Within 3 months of condition
  The number of living donors screened on behalf of transplant candidates will be collected/ identified through the electronic medical record system.
Number of Live Donor Approvals | Within 3 months of condition
  The number of living donor approvals on behalf of transplant candidates will be collected/ identified through the electronic medical record system.

CONTACTS AND LOCATIONS:
Overall Officials: Vineeta Kumar, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No